CLINICAL TRIAL: NCT00511654
Title: A Parallel Group, Single-Blind, Randomised, Placebo Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GW823296 and Its Effect on the Pharmacokinetics of Midazolam After Once-Daily Repeated Oral Doses in Healthy Subjects
Brief Title: 28-day Repeat Dose and Drug Interaction Study With Orvepitant (GW823296)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: NKG10004
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Depressive Disorder
Keywords: depression; NK1 receptor antagonists,
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — orvepitant; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects in Group 1 receiving GW823296 (Experimental): Subjects will receive single dose of GW823296 on Day 1 followed by a wash-out period of 1 week. The subjects will then be administered GW823296 for 28 days in the repeat dosing period.
  Interventions: Drug: GW823296 tablet
- Subjects in Group 1 receiving placebo (Placebo Comparator): Subjects will receive single dose of placebo on Day 1 followed by a wash-out period of 1 week. The subjects will then be administered placebo for 28 days in the repeat dosing period.
  Interventions: Drug: GW823296 matching placebo
- Subjects in Group 2 and 3 receiving GW823296 (Experimental): Subjects will receive single dose of midazolam on Day 1 followed by wash-out period of one day. Further the subjects will be administered GW823296 on Day 3 of single dose period followed by a wash-out period of 1 week. The subjects will then be administered a single dose of GW823296 for 28 days (Day 1 to Day 28 of repeat dosing period) and a single dose of midazolam on Day 29 of repeat dosing period.
  Interventions: Drug: GW823296 tablet; Drug: Midazolam
- Subjects in Group 2 and 3 receiving placebo (Placebo Comparator): Subjects will receive single dose of midazolam on Day 1 followed by wash-out period of one day. Further the subjects will be administered placebo on Day 3 of single dose period followed by a wash-out period of 1 week. The subjects will then be administered a single dose of placebo for 28 days (Day 1 to Day 28 of repeat dosing period) and a single dose of midazolam on Day 29 of repeat dosing period.
  Interventions: Drug: GW823296 matching placebo; Drug: Midazolam

INTERVENTIONS:
Drug: GW823296 tablet — GW823296 immediate release tablets will be available as white film-coated tablets containing 5 milligrams (mg) and 20 mg of GW823296 for oral administration.
  Other Names: Orvepitant
  Arms: Subjects in Group 1 receiving GW823296; Subjects in Group 2 and 3 receiving GW823296
Drug: GW823296 matching placebo — Matching placebo tablets will be identical in appearance to the GW823296 tablets.
  Arms: Subjects in Group 1 receiving placebo; Subjects in Group 2 and 3 receiving placebo
Drug: Midazolam — Midazolam will be administered as 5 milliliter (mL) of an intravenous solution for oral application (5 mg/5 mL, Dormicum).
  Arms: Subjects in Group 2 and 3 receiving GW823296; Subjects in Group 2 and 3 receiving placebo

SUMMARY:
This study is being conducted to obtain information on the safety and tolerability of repeated doses of GW823296 for 28 days in healthy male and female subjects. In addition, the pharmacokinetics of GW823296 will be evaluated to confirm the doses to be used in Phase II efficacy studies. The effect of repeat dose (RD) of GW823296 on CYP3A4 enzyme activity will be investigated evaluating the pharmacokinetics of midazolam and urine 6-?-hydroxycortisol/cortisol ratio.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a Physician Responsible, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring. A subject with a clinical abnormality or laboratory variables outside the reference range for the population being studied, with the exception of liver transaminases, troponin I and TSH, may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures. Please note that subjects should have liver transaminases, troponin I and TSH values within the range specified in the exclusion criteria below.
* Women of non-childbearing potential (i.e., physiologically incapable of becoming pregnant with documentation of hysterectomy or bilateral ovariectomy >6 months, including any female who is postmenopausal. For purposes of this study, postmenopausal is defined as one year without menses and confirmed by FSH according to the local laboratory ranges at screening) and having a negative serum hCG pregnancy test at screening.
* No co-morbid Psychiatric Disorders as defined using the Mini International Neuropsychiatric Interview (M.I.N.I) scale
* Aged 18-65 years, inclusive
* A 12-lead ECG and 24-hours Holter ECG at screening showed no abnormalities that in the opinion of the Principal Investigator will compromise safety in this study
* Body weight >50 kg and body mass index (BMI) within the range 19.0-29.9 kg/m2
* Subjects with a history of peptic ulcer disease (PUD) with a known aetiology must provide documentation by a gastroenterologist of the aetiology of the PUD and that effective treatment was provided with full eradication of ulcers and symptoms. For such subjects appropriate steps must also have been taken to minimize reoccurrence risk (i.e. if PUD was nonsteroidal anti-inflammatory drug [NSAID] induced, the subject should no longer be taking NSAID medications; if cause was Helicobacter pylori [H. pylori], the subject should have been appropriately treated). For all subjects, regardless of whether there is a positive history of PUD, sites are required to document their H. pylori status at screening. Entry into the study is permitted for subjects who are seropositive for H. pylori, but treatment is recommended, either before or after study participation at the discretion of the Principal Investigator.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* The subject must be able to read, comprehend and record information.
* A signed and dated written informed consent is obtained from the subject.
* The subject is available to complete the study.

Exclusion Criteria:

* The subject has screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5x upper limit of the normal range (ULN); testing may be repeated once to see if value returns to within acceptance range but any such laboratory abnormality must be resolved by the baseline visit.
* Subjects with a troponin I value >0.032 ng/mL at screening are not eligible. Testing may not be repeated. The subject should be referred to the treating physician for further evaluation, as appropriate.
* Subjects with a TSH value above the upper limit of the normal range (ULN) at screening are not eligible. The subject should be referred to the treating physician for further evaluation, as appropriate. Testing may be repeated once to see whether the value returns to within normal range but such abnormality must be resolved before the baseline visit.
* Subjects found to have stool positive for occult blood. If such a stool was obtained without the subject abstaining from red meat for 3 or more days prior to testing, this may be repeated once following such abstinence. If that stool is negative for occult blood the subject is considered eligible.
* Subjects with known or suspected iron deficiency
* Subjects with a history of myopathy or rhabdomyolysis
* The subject is unable to abstain from strenuous physical activity for 72 hours prior to screening, for 72 hours prior first dosing until the last PK sample has been collected, and for 72 hours prior to the follow-up visit.
* The subject has donated a unit of blood (450 mL) within the previous 60 days or intends to donate in the month after completing the study.
* The subjects is currently taking regular (or a course of) medication whether prescribed or not, including vitamins and herbal remedies, such as St John's Wort. Any concurrent medication will not be permitted for 48 hours before admission to the CPRU until the end of the study period (follow-up visit).
* Typical consumption of more than 14 alcoholic units in any week, or more than 3 (for males) or 2 (for females) alcoholic units in any single day, over the month preceding the screening visit [NOTE: 1 unit = 8 oz beer, 3 oz wine, or 1 oz hard liquor]
* The subject smokes or has smoked in the last 3 months.
* The subject has tested positive for Hepatitis C antibody or Hepatitis B surface antigen.
* The subject has tested positive for HIV-1/2.
* The subject has a past history of drug abuse or has tested positive for urine drugs of abuse at screening. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.
* Male subject intends to father a child during the study and the 3 months following the study
* Subjects with a history of eye disease (excluding moderate myopia) or clinically relevant eye examination finding, which in the opinion of the study ophthalmologist contraindicates their participation in the study
* Vulnerable subject (e.g. kept in detention)
* Subjects who have had hypersensitivity or intolerance to NK1 antagonists
* Subject has a known hypersensitivity against midazolam or against one of the excipients of Dormicum® (subjects of Cohorts 2 and 3 only)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-06-12 (Actual); Primary Completion 2008-01-11 (Actual); Study Completion 2008-01-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of oral doses of GW823296 given once daily for 28 days in healthy male and female subjects | Up to Day 43

SECONDARY OUTCOMES:
To assess the PK of single oral doses of GW823296 given once daily for 28 days and its potential to alter the CYP3A4 enzyme activity in healthy male and female subjects. Pharmacogenetics. | Up to Day 31
PK parameters of GW823296 following repeated oral doses of the GW823296 given once daily: Cmax, tmax, AUC0-τ, accumulation ratio (Ro) and, if possible, lz, t1/2,z, and time invariance (Rs) | Up to Day 31
Effect of repeated daily oral doses of GW823296 on the PK of single doses of midazolam: Cmax, tmax, AUC0-t, and, if possible, AUC0-∞ and lz and t1/2,z of midazolam | Up to Day 30
Effect of repeated daily oral doses of GW823296 on urine 6-b-hydroxycortisol / cortisol ratio | Up to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- See also: Results for study NKG10004 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/NKG10004?search=study&search_terms=NKG10004#rs